CLINICAL TRIAL: NCT02693756
Title: Home-based Motor Imagery Intervention for the Improvement of Gait Stability in Elderly Persons. A Cross-over Feasibility Study.
Brief Title: Home-based Motor Imagery for Gait Stability in Older Adults. A Cross-over Feasibility Study. (MIGS-F)
Acronym: MIGS-F
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Principal Investigator, Roger Hilfiker, Prof. Roger Hilfiker, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PHYVS2016-1
Record Dates: First submitted 2016-02-07; First posted 2016-02-29 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Gait, Unsteady
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants will be allowed to perform all usual activities but should refrain from performing the motor imagery exercises.
- Motor imagery (Experimental): The motor imagery intervention is a non-pharmacological and non-invasive treatment often used in sport, music, or physical rehabilitation (Schuster, Hilfiker et al. 2011). Proposed tasks to be imagined by the participants are for example:
  "Imagine you are walking on ice. During the first steps, you are slipping quite often, but as you walk on, your steps become more stable and you walk without problems over the ice. Try to imagine how you react when you slip on ice, how you try not to fall and to continue to walk normally" The motor imagery intervention will be performed independently by the study participants at home without supervision three times a week for three weeks.
  Interventions: Other: Motor imagery

INTERVENTIONS:
Other: Motor imagery — The motor imagery intervention is a non-pharmacological and non-invasive treatment often used in sport, music, or physical rehabilitation (Schuster, Hilfiker et al. 2011). Proposed tasks to be imagined by the participants are for example:
  "Imagine you are walking on ice. During the first steps, you are slipping quite often, but as you walk on, your steps become more stable and you walk without problems over the ice. Try to imagine how you react when you slip on ice, how you try not to fall and to continue to walk normally" The motor imagery intervention will be performed independently by the study participants at home without supervision three times a week for three weeks.
  Arms: Motor imagery

SUMMARY:
Gait stability is reduced as early as from age 40 to 50. Gait stability can be improved in patients with neurological diseases or in healthy elderly persons with exercises.

There is evidence that mental practice, also called motor imagery, the imagination of performing a movement, can also improve an activity or balance. The effective performance and the imagination of a task activates some overlapping central areas and neural networks, which might explain the improvements after motor imagery.

The investigators set out to test the feasibility of such a study using an open label randomized cross-over trial including 32 persons aged 40 years or more. The primary aim is to evaluate whether the instructions are clear, the intervention and the study procedures are acceptable and to assess the proportion of participants withdraw from the study (drop outs). Secondary aims are the assessment of between group differences in the changes of the gait stability.

DETAILED DESCRIPTION:
Gait stability is reduced as early as from age 40 to 50. Gait stability can be improved in patients with neurological diseases or in healthy elderly persons with exercises.

There is evidence that mental practice, also called motor imagery, the imagination of performing a movement, can also improve an activity or balance. The effective performance and the imagination of a task activates some overlapping central areas and neural networks, which might explain the improvements after motor imagery.

These "non-physical kind of training" modalities could be used in patients who are immobilized temporarily (bedridden because of non-chronic disease, infection etc.), or in those who are not allowed to charge their leg normally (e.g. postoperative phase of joint replacement or fractures), or it can be used in combination with physical exercises, or in the preparation of the physical exercise training (either skilling up phase or as a preparation to increase safety of physical exercises). In persons above 40 years of age, motor imagery could provide a sound exercise modality for tasks that are not easy to perform with real performance. For example, walking on slippery underground such as ice, walking on a small trail in some altitude, avoiding running dogs or cats on a sidewalk, or catching up after stumbling can be either difficult to exercise in reality or might be too dangerous in reality. Imaging one's performance in such difficult environments or situations might lead to better gait stability, improved reactions in these situations and thus probably to reduced falls frequency.

Gait stability can be estimated with the local dynamic stability, which is based on chaos theory, i.e. the maximal Lyapunov exponent, is strongly influenced by the sensorimotor balance system and is widely used for measuring gait stability.

In the future, the investigators plan a large scale randomized open label cross-over study to test whether nine sessions of motor imagery improve walking stability, measured with the Lyapunov Exponent.

To prepare this future study, the investigators set out to test the feasibility of such a study with a feasibility study using an open label randomized cross-over trial including 32 persons aged 40 years or more. The primary aim is to evaluate whether the instructions are clear, the intervention and the study procedures are acceptable and to assess the proportion of participants withdraw from the study (drop outs). Secondary aims are the assessment of between group differences in the changes of the gait stability.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old or older
* Able to walk bout 100 meter, with or without walking aids, but without the help of a person or an ambulator

Exclusion Criteria:

* Walking with an ambulator (Rollator)
* No able to understand German

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-02; Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint "feasibility" | Immediately after the end of the both Intervention periods (week 6)
  Combination of the following three parts:
  Part 1: one question about the understandability of the exercises Part 2: one question about the acceptability of the whole study process Part 3: Finishing the whole study: Did the participant finish the whole study, i.e. all three test sessions and at least some session of motor imagery exercises (based on the exercise calendar)?

SECONDARY OUTCOMES:
Adherence to the motor imagery exercises | Immediately after the end of the first intervention periods (week 3)
  The adherence to the motor imagery exercises will be assessed with a exercise calendar with a sheet for each of the three weeks. On each day of the calendar the exercises were shortly described and the participants can just check whether he has done that exercise and can state how many minute he or she has exercises that day (only motor imagery exercises).
Change in the Lyapunov Exponent in the three acceleration axes "anterio-posterior", "medio-lateral" and "vertical" | Immediately after the end of the first period (week 3)
  The "first" endpoint for effectiveness is the change in the Lyapunov Exponent in the three acceleration axes "anterio-posterior", "medio-lateral" and "vertical". The Lyapunov Exponent is calculated based on the 4 times 30 meter walk test in normal speed.
  For these tests, the participants wear normal clothes and normal shoes (same shoes at all three test sessions). The test will be performed in a 35 meter long corridor.
  The participant starts walking with his normal speed, walks 30 meters and stops. He turns 180°, waits ten seconds and starts walking again the 30 meters. He repeats this until he has four series of 30 meters. The data will be stored after each participant on a portable computer in coded form. The Lyapunov Exponent is then calculated later in R (statistical software) and the mean over all four series is taken.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Hilfiker, Principal Investigator — School of Health Sciences, HES-SO Valais-Wallis
Locations (1):
- Hochschule für Gesundheit HES-SO Valais-Wallis, Leukerbad, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: No